CLINICAL TRIAL: NCT06721624
Title: Prospective Observational Study of Naturopathic Approaches to IBS
Status: Recruiting | Type: Observational
Sponsor: National University of Natural Medicine (Other)
Collaborators: Gastroenterology Association of Naturopathic Physicians (Unknown)
Responsible Party: Sponsor
Other Study IDs: RB82224
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Irritable Bowel Syndrome; IBS; naturopathy; naturopathic medicine
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Naturopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Naturopathic medicine — Whole system naturopathic medicine

SUMMARY:
Irritable bowel syndrome (IBS) is a common condition affecting about 4% of people worldwide and can significantly impact quality of life and healthcare costs. While there are medications available, few are consistently effective, leading many people with IBS to explore alternative treatments, including naturopathy. However, research on naturopathic approaches to IBS is limited.

This study aims to describe how naturopathy is used to treat IBS and to collect preliminary data on changes in IBS symptoms before and after treatment. It will use a prospective, observational design without a control group, focusing on outcomes from individualized naturopathic care provided by licensed practitioners.

Adult patients with diagnosed IBS or IBS-like symptoms will be recruited from naturopathic doctors affiliated with the Gastroenterology Association of Naturopathic Physicians. Participants' IBS symptoms will be assessed using validated tools (IBS-SSS and IBS-AR), and quality of life will be measured using the PROMIS-29 survey. Treatment details and any adverse effects will also be recorded. The main outcome will be the difference in symptoms and quality of life after 12 weeks of treatment. Results will be analyzed with statistical tests (p-value < 0.05) and summarized.

The findings from this pilot study will help fill knowledge gaps and provide a foundation for designing a more rigorous randomized controlled trial in the future.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common functional bowel disorder with a worldwide prevalence of about 4% according to the Rome IV criteria. It has a significant impact on quality of life and societal expense. While there are pharmaceutical options available, few can be reliably recommended. Many IBS sufferers turn to complementary and alternative medicine, including naturopathy. Naturopathic approaches to IBS are poorly studied to date. The researchers aim to describe naturopathic approaches to IBS, as well as establish pilot data on before-and-after changes in validated IBS instruments. The study will employ a prospective, observational, naturalistic design. The uncontrolled before-and-after study will examine the outcomes associated with individualized, whole system naturopathic care as determined by each respective provider. The researchers will recruit adult patients either diagnosed with IBS or presenting with IBS-like symptoms, and presenting to the private practices of naturopathic doctors who are members of the Gastroenterology Association of Naturopathic Physicians. Participants' IBS symptoms will be measured using validated instruments (IBS-SSS and IBS-AR). Quality of life will be measured by the PROMIS - 29. Adverse events will be tracked, as will treatment descriptions. The primary outcomes will be before-and-after differences using week 12 as the primary endpoint. P-values will be set at 0.05 and descriptive and summary data will be presented. This study is designed to contribute to significant evidence gaps and to gather preliminary evidence to guide the design of a follow-up randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) who present with a pre-existing IBS diagnosis or IBS- like gastrointestinal symptoms.
* Pre-existing IBS diagnosis or IBS-like gastrointestinal symptoms must be the primary cause of the visit.
* An IBS diagnosis must be listed within the top 3 diagnoses for the visit and addressed in the individualized treatment plan.

Exclusion Criteria:

*Inability to read and write in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are adults (≥18 years of age) who present to the clinical co-investigators' practices with a pre-existing IBS diagnosis (or IBS-like gastrointestinal symptoms which lead to clinical personnel making a diagnosis of IBS via Rome IV criteria) as the primary cause of their visit.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
IBS Severity | 6 months
  IBS-SSS
Health Status | 6 months
  PROMIS-29

SECONDARY OUTCOMES:
Adequate Relief | 6 months
  IBS-AR
CARE | 6 months
  The clinician's interpersonal practice will be described primarily through the CARE measure, a 10-item validated instrument designed to evaluate patient experiences of practitioner empathy. The CARE measure has demonstrated validity across a variety of health-care settings and its preliminary application in CIH settings suggests reliability in this setting
Patient empowerment | 6 months
  The 5-item Empowerment scale will be employed to evaluate the patient experiences of the clinical consultation with regards to the degree to which the practitioner encourages patient empowerment.
The Patient-Centered Care-Perceived Provider Support-Empowerment Scale | 6 months
  The Patient-Centered Care-Perceived Provider Support-Empowerment Scale is a trifecta of validated instruments developed to assess patients' perceptions of provider support, patient-centered care, and empowerment as they relate to health outcomes. These questionnaires aim at measuring the impact of the therapeutic relationship, the philosophy of healing, and CIH-specific techniques on treatment effects.
Diagnosis and treatment characteristics | 6 months
  The naturopathic diagnosis and treatment characteristics for each participant will also be extracted from patient charts. In particular, the naturopathic and differential diagnosis, and details of all prescribed treatments (e.g. diets, supplements, medications, lifestyle changes), including doses and frequencies.
Adverse Events | 6 months
  Total number of adverse events and serious adverse events (using NIH's Common Terminology Criteria for Adverse Events version 4.0). This will be measured by practitioner report using chart abstraction. Practitioners will be trained on grading and documenting adverse events, as well as using standardized AE forms, before subjects are enrolled.

CONTACTS AND LOCATIONS:
Locations (1):
- Helfgott Research Institute - National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided